CLINICAL TRIAL: NCT01778972
Title: Fall Prevention for Old Community-dwelling People in Uppsala, Västerås and Sörmland
Brief Title: Fall Prevention for Old Community-dwelling People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, karin hellstrom, PhD, Senior Lecturer, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fall prevention UV; 307301 (Other Grant/Funding Number: Regional forskningsrådet i Uppsala- och Örebroregionen)
Record Dates: First submitted 2013-01-16; First posted 2013-01-29 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2019-04

CONDITIONS: Physical Activity
Keywords: Fall prevention; Home exercise; Strength training; Balance training
MeSH Terms: conditions — Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Otago home training programme (Experimental): Otago home exercise programme was designed specifically to prevent fall. It consists of a set of leg muscle strengthening and balance retraining exercises progressing in difficulty, and a walking plan.
  The exercise are individually prescribed and increase in difficulty during a series of five home visits by a physiotherapist.
  Interventions: Other: Otago home exercise programme
- Motivational interviewing plus Otago (Experimental): This group is not only exercising at home but also getting motivational interviewing from the physiotherapist at he five home visits. The physiotherapists doing motivational interviewing are specially trained in motivational interviewing.
  Interventions: Other: Motivational interviewing plus Otago
- Control grop (No Intervention): Participants are instructed to live their ordinary lives.

INTERVENTIONS:
Other: Otago home exercise programme — Otago home exercise program was designed specifically to prevent falls. It consists of a set of leg muscle strengthening and balance retraining exercises progressing in difficulty, and a walking plan.
  The exercise are individually prescribed and increase in difficulty during a series of five home visits by a physiotherapist.
  Arms: Otago home training programme
Other: Motivational interviewing plus Otago — This group is not only exercising at home but also getting motivational interviewing from the physiotherapist at he five home visits. The physiotherapists doing motivational interviewing are specially trained in motivational interviewing.
  Arms: Motivational interviewing plus Otago

SUMMARY:
Fall-related injuries are a major health problem in the growing older population. Most older people are not aware of that physical training can decrease the risk of falling. The aim of tha study is to investigate the effect of the Otago home exercise programme with and without motivational interviewing in community-dwelling people 75 years or older on frequence of falls, fall-related injuries, physical capacity, fall-related self-efficacy, quality of life, mortality and health-related costs.

DETAILED DESCRIPTION:
Participants in the two intervention groups will exercise at home with supervision from physiotherapist week one, two, four and eight. They will then be contacted for telephone follow-up month five, seven and twelve after the start of training. The control group is encouraged to live as usual.

All participants are assessed at baseline, after three, 12 and 24 months from inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

75 years or older, community-dwelling, in need of homecare or rollator

Exclusion Criteria:

Cognitive impairment (below 25 on Mini Mental test) Not able to transfer independently indoors -

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2012-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Frequence of falls will be measured with a monthly fall-calender | Two year
  A fall-calender with registration of falls on a monthly bases will be used to record falls. The fall-calender should be sent in each month. Falls will be followed-up with telephone interviews.

SECONDARY OUTCOMES:
Fall-related injuries will be measured by telephone interviews. | Two years
Physical performance will be measured with Short Physical Performance Battery (SPPB) | Two years
  SPPB measures balance, functional leg strength and walking speed.
Dynamic balance will be assessed with Mini-BESTest | Two years
  Mini-BESTest assess dynamic balance impairments in 14 items. The items covers a broad spectrum of performance tasks, including transitions and anticipatory postural adjustments, postural responses to to perturbation, sensory orientation and dynamic stability in gait.

OTHER OUTCOMES:
Fall-related self-efficacy will be measured with Fall efficacy scale, Swedish version. | Two years
Grip strength will be measured with Jamar Hand Dynamometer | Two years
Physical Activity level will be measured with Frändin/Grimby activity scale. | Two years
Health related quality of life will be measured with European quality of life questionaire (EQ-5D). | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Karin E Hellström, PhD, Principal Investigator — Uppsala University; Ann-Christin Johansson, PhD, Principal Investigator — Mälardalens University, Sweden; Anne Söderlund, Professor, Principal Investigator — Mälardalens University, Sweden
Locations (2):
- Sweden (2):
  - Homes, Uppsala
  - Homes, Västerås

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- [Derived] Arkkukangas M, Hultgren S. Implementation of motivational interviewing in a fall prevention exercise program: experiences from a randomized controlled trial. BMC Res Notes. 2019 May 14;12(1):270. doi: 10.1186/s13104-019-4309-x. PMID 31088557